CLINICAL TRIAL: NCT01169779
Title: Efficacy and Safety of Lixisenatide in Patients With Type 2 Diabetes Mellitus Insufficiently Controlled by Metformin (With or Without Sulfonylurea): a Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study With 24-week Treatment Period
Brief Title: Efficacy and Safety of Lixisenatide in Patients With Type 2 Diabetes Mellitus Insufficiently Controlled by Metformin
Acronym: GetGoal-M-Asia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC11321; U1111-1116-8938 (Other: UTN)
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 1-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 2 weeks, followed by 20 mcg QD up to Week 24.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin; Drug: Sulfonylurea
- Placebo (Placebo Comparator): 1-step initiation regimen of volume matching placebo: 10 mcg QD for 2 weeks, followed by 20 mcg QD up to Week 24.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Metformin; Drug: Sulfonylurea

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Placebo — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Metformin — Metformin to be continued at stable dose (at least 1.0 gram per day and not more than 1.5 gram per day) up to Week 24.
Drug: Sulfonylurea — Sulfonylurea if given at screening, to be continued up to Week 24. In patients with a screening HbA1c <8% the dose is decreased by 25% to 50% at randomization and then increased up to the screening dose between Week 4 and 12 as per fasting self-monitored plasma glucose (SMPG) values. In patients with a screening HbA1c >=8%, the dose is not to be changed at randomization. In any case, after Week 12, sulfonylurea is to be continued at a stable dose.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010) in comparison to placebo, as an add-on treatment to metformin with or without sulfonylurea, over a period of 24 weeks of treatment.

The primary objective is to assess the effects on glycemic control of lixisenatide (AVE0010) in comparison to placebo as an add-on treatment to metformin with or without sulfonylurea in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 24.

The secondary objectives are to assess the effects of lixisenatide over 24 weeks on percentage of patients reaching HbA1c less than (< ) 7 percent (%) or HbA1c less than or equal to (<=) 6.5%, fasting plasma glucose (FPG), 2-hour postprandial plasma glucose (PPG) and glucose excursion during standardized meal test, body weight; to evaluate safety, tolerability, pharmacokinetic (PK) and anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
The study duration for each patient is 27 weeks +/- 10 days (up to 2 weeks screening + 1 week run-in + 24 weeks double-blind treatment + 3 days follow-up).

ELIGIBILITY:
Inclusion criteria:

- Type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit, insufficiently controlled with metformin alone or metformin with sulfonylurea at the time of the screening visit

Exclusion criteria:

* HbA1c <7% or greater than (>) 10% at screening
* At the time of screening age < legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Treatment with metformin not at a stable dose of at least 1.0 gram per day or more than 1.5 gram per day for at least 3 months prior to screening visit
* In case of treatment with sulfonylurea, if the sulfonylurea dosage is less than the maximum effective dose (that is, half of the maximum recommended dose according to local labeling), or is not at a stable (unchanged) dose for at least 3 months prior to screening
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* History of hypoglycemia unawareness
* Body mass index <=20 kilogram per square meter (kg/m^2)
* Weight change of >5 kg during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, or inflammatory bowel disease or patients considered by the investigator at high risk for acute pancreatitis (for example, with known history of biliary gallstone[s], or with very high triglyceride level [>=5.65 mmol/L]) at the time of screening
* Personal or family history of medullary thyroid cancer or genetic conditions that predispose to medullary thyroid cancer (for example, multiple endocrine neoplasia syndromes);
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure (SBP) or diastolic blood pressure (DBP) >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: amylase and/or lipase: >3 times upper limit of normal (ULN); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; calcitonin >20 picogram per milliliter (5.9 picomole per liter) ; and positive test for Hepatitis B surface antigen and/or Hepatitis C antibody
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram, or vital signs at the time of screening that, in the judgment of the investigator or any sub-investigator, precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as attending scheduled visits, being able to do self-injections; likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol; investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of oral or injectable antidiabetic or hypoglycemic agents other than metformin and sulfonylurea (for example, alpha-glucosidase inhibitor, thiazolidinedione, glucagon-like peptide -1 [GLP-1], receptor agonist, dipeptidyl-peptidase-4 inhibitors, insulin) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to screening;
* Participation in a previous study with lixisenatide
* Renal impairment defined with creatinine >1.4 mg/dL in women and creatinine >1.5 mg/dL in men
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis, unstable (that is, worsening) and not controlled (that is, prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any GLP-1 agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (35):
- China (28):
  - Investigational Site Number 156011, Beijing
  - Investigational Site Number 156012, Beijing
  - Investigational Site Number 156019, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156003, Beijing
  - Investigational Site Number 156009, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156036, Changchun
  - Investigational Site Number 156016, Changsha
  - Investigational Site Number 156015, Changsha
  - Investigational Site Number 156006, Chengdu
  - Investigational Site Number 156032, Chengdu
  - Investigational Site Number 156010, Dalian
  - Investigational Site Number 156004, Guangzhou
  - Investigational Site Number 156008, Guangzhou
  - Investigational Site Number 156025, Guangzhou
  - Investigational Site Number 156031, Haikou
  - Investigational Site Number 156014, Harbin
  - Investigational Site Number 156029, Hefei
  - Investigational Site Number 156013, Qingdao
  - Investigational Site Number 156007, Shanghai
  - Investigational Site Number 156030, Shanghai
  - Investigational Site Number 156020, Shenyang
  - Investigational Site Number 156035, Suzhou
  - Investigational Site Number 156033, Taiyuan
  - Investigational Site Number 156037, Tianjin
  - Investigational Site Number 156022, Xi'an
  - Investigational Site Number 156023, Xi'an
- Hong Kong (3):
  - Investigational Site Number 344001, Hong Kong
  - Investigational Site Number 344003, Hong Kong
  - Investigational Site Number 344002, Shatin, Nt
- Malaysia (3):
  - Investigational Site Number 458001, Kelantan
  - Investigational Site Number 458003, Kuala Lumpur
  - Investigational Site Number 458002, Putrajaya
- Investigational Site Number 764002, Bangkok, Thailand

REFERENCES:
- [Result] Yu Pan C, Han P, Liu X, Yan S, Feng P, Zhou Z, Lv X, Tian H, Jin Kui Y, Su B, Shang S, Niemoeller E. Lixisenatide treatment improves glycaemic control in Asian patients with type 2 diabetes mellitus inadequately controlled on metformin with or without sulfonylurea: a randomized, double-blind, placebo-controlled, 24-week trial (GetGoal-M-Asia). Diabetes Metab Res Rev. 2014 Nov;30(8):726-35. doi: 10.1002/dmrr.2541. PMID 24639432
- [Derived] Seino H, Onishi Y, Naito Y, Komatsu M. Lixisenatide improves glycemic outcomes of Japanese patients with type 2 diabetes: a meta-analysis. Diabetol Metab Syndr. 2016 Jun 1;8:36. doi: 10.1186/s13098-016-0151-7. eCollection 2016. PMID 27252787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 centers in 4 countries between July 21, 2010 and December 22, 2011.
Pre-assignment Details: A total of 655 patients were screened of which 264 (40.3%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 391 patients were randomized.
Groups:
- Placebo: 1-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 2 weeks, followed by 20 mcg QD up to Week 24.
- Lixisenatide: 1-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 2 weeks, followed by 20 mcg QD up to Week 24.
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 195 (Randomized.) | 196
Treated/Safety Population | 194 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 196
Modified Intent-to-Treat(mITT)Population | 193 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 195
Subgroup for Standardized Meal Test | 130 (Patients at selected sites where standardized meal test was performed.) | 121
Completed | 184 | 179
Not Completed | 11 | 17
Not completed — Adverse Event | 3 | 11
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Familial and personal reasons | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo: 1-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 2 weeks, followed by 20 mcg QD up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 194 | 196 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.5) | 54.5 (10.3) | 54.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 95 | 198
  Male | 91 | 101 | 192
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Asian/Oriental | 194 | 196 | 390
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.85 (0.71) | 7.95 (0.81) | 7.90 (0.76)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 8.74 (1.83) | 8.84 (2.12) | 8.79 (1.98)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients analyzed = 130 and 121 for Placebo and Lixisenatide treatment arm, respectively, as meal challenge test was performed at selected sites only.
  mmol/L | 17.19 (4.06) | 16.07 (3.77) | 16.65 (3.95)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients analyzed = 130 and 121 for Placebo and Lixisenatide treatment arm, respectively, as meal challenge test was performed at selected sites only.
  mmol/L | 8.14 (3.11) | 7.12 (3.21) | 7.65 (3.20)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 72.74 (13.64) | 73.18 (13.93) | 72.96 (13.77)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.84 (4.80) | 6.45 (4.64) | 6.64 (4.72)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 27.08 (3.75) | 26.75 (3.86) | 26.91 (3.80)
Metformin Daily Dose [Mean (Standard Deviation); unit: milligram (mg) per day] | 1363.4 (221.9) | 1369.9 (219.9) | 1366.7 (220.7)
Number of Patients With Sulfonylurea use at Baseline [Number; unit: participants]
  Yes | 92 | 82 | 174
  No | 102 | 114 | 216

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline on-treatment assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo: 1-step initiation regimen of volume matching placebo.
- Lixisenatide: 1-step initiation regimen of lixisenatide.
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 188 | 185
percentage of hemoglobin | -0.47 (0.104) | -0.83 (0.102)
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; To detect a difference of 0.5% in change in HbA1c at Week 24 between lixisenatide arm and placebo arm, 190 patients per group would provide a power of 96% assuming common standard deviation of 1.3% with 2-sided test at 5% significance level; Test type: Superiority or Other; p = 0.0004, ANCOVA — Statistical testing:2-sided at significance level=0.05. Analysis of co-variance (ANCOVA) included treatment arms, randomization strata of screening HbA1c (<8.0,>=8.0%), sulfonylurea use (Yes,No), country as fixed effects, baseline HbA1c as covariate; Least squares (LS) mean difference = -0.36, 95% CI 2-sided [-0.551 to -0.162], Standard Error of Mean 0.099

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting Baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 1 day after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline on-treatment assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 191 | 190
mmol/L | -0.21 (0.200) | -0.69 (0.197)

3. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change was calculated by subtracting Baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 116 | 107
mmol/L | -1.33 (0.376) | -5.61 (0.393)

4. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting Baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline on-treatment assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 191 | 188
kilogram | -1.24 (0.273) | -1.50 (0.267)

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline on-treatment assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 188 | 185
percentage of participants | 38.8 | 53.0

6. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 5
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 188 | 185
percentage of participants | 18.1 | 32.4

7. Secondary Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change was calculated by subtracting Baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with Baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 116 | 106
mmol/L | -0.79 (0.340) | -4.78 (0.356)

8. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 5
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 191 | 188
percentage of participants | 14.7 | 19.7

9. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During Main 24-Week Period
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >250 milligram/deciliter (mg/dL) (13.9 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >220 mg/dL (12.2 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline on-treatment assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 193 | 195
percentage of participants | 6.7 | 3.6

10. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 194 | 196
participants
  Symptomatic hypoglycemia | 5 | 11
  Severe symptomatic hypoglycemia | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration
Description: Median exposure to study treatment was 169 days for both treatment arms. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 4/194 | 3/196
Other Adverse Events (participants affected / at risk) | 46/194 | 80/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=194) | Lixisenatide (N=196)
Anaphylactic shock (Immune system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=194) | Lixisenatide (N=196)
Upper respiratory tract infection (Infections and infestations) | 8 | 12
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 18 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 8 | 17
Nausea (Gastrointestinal disorders) | 5 | 32
Vomiting (Gastrointestinal disorders) | 2 | 15
Diabetic nephropathy (Renal and urinary disorders) | 13 | 13
Blood glucose decreased (Investigations) | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.